CLINICAL TRIAL: NCT02745860
Title: Single-center, Open-label, Randomized, Two-way Crossover Study in Healthy Adult Male Subjects to Compare the Pharmacokinetics of Selexipag (ACT-293987) Following Single Oral Administration of 4 Film-coated Pediatric Tablets of 50 µg vs One Film-coated Tablet of 200 µg Selexipag
Brief Title: Comparison of Two Dose Strengths of Selexipag in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AC-065-112
Record Dates: First submitted 2016-04-18; First posted 2016-04-20 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy Subjects
Keywords: selexipag; pharmacokinetics
MeSH Terms: interventions — selexipag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence AB (Experimental): Subjects receive 200 µg of selexipag (adult formulation) as a single oral dose during Period 1 and 200 µg of selexipag (pediatric formulation) as a single oral dose during Period 2
  Interventions: Drug: Selexipag (adult formulation); Drug: Selexipag (pediatric formulation)
- Sequence BA (Experimental): Subjects receive 200 µg of selexipag (pediatric formulation) as a single oral dose during Period 1 and 200 µg of selexipag (adult formulation) as a single oral dose during Period 2
  Interventions: Drug: Selexipag (adult formulation); Drug: Selexipag (pediatric formulation)

INTERVENTIONS:
Drug: Selexipag (adult formulation) — One selexipag film-coated tablet of 200 µg
  Other Names: ACT-293987
Drug: Selexipag (pediatric formulation) — Four selexipag film-coated tablets of 50 µg
  Other Names: ACT-293987

SUMMARY:
Clinical study in healthy adult subjects to compare the adult tablet of selexipag with the tablet developed for children.

DETAILED DESCRIPTION:
Healthy male adults receive a single dose of selexipag (200 µg) but using a different tablet strength (4 film-coated pediatric tablets of 50 µg versus one film-coated tablet of 200 µg selexipag) during each of the two study periods. There is a washout of 7-9 days between the two study treatment administrations.

ELIGIBILITY:
Key inclusion Criteria:

* Male subjects aged from 18 to 45 years (inclusive) at screening
* Signed informed consent form
* Body mass index (BMI) between 18.0 and 28.0 kg/m2 (inclusive) at screening
* Healthy on the basis of physical examination,cardiovascular assessments and laboratory tests

Key exclusion Criteria:

* Any contraindication to the study treatments
* History or clinical evidence of any disease or medical / surgical condition or treatment, which may put the subject at risk of participation in the study or may interfere with the absorption, distribution, metabolism or excretion of the study treatments
* Any circumstances or conditions, which, in the opinion of the investigator, may affect the subject's full participation in the study or compliance with the protocol

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve [AUC(0-inf)] of selexipag and ACT-333679 | From predose until 72 hours postdose for each treatment period
  AUC(0-inf) is the area under plasma concentration-time curves for selexipag and its metabolite (ACT-333679), calculated from zero to the extrapolated infinite time
Maximum plasma concentration (Cmax) of selexipag and ACT-333679 | From predose until 72 hours postdose for each treatment period
  Cmax is directly derived from the individual plasma concentration time curves for selexipag and its metabolite ACT-333679

SECONDARY OUTCOMES:
Time to reach Cmax (tmax) of selexipag and ACT-333679 | From predose until 72 hours postdose for each treatment period
  tmax is directly derived from the individual plasma concentration time curves for selexipag and its metabolite ACT-333679
Terminal half-life (t½) of selexipag and ACT-333679 | From predose until 72 hours postdose for each treatment period
  The period of time required for the concentration levels of selexipag or its metabolite (ACT-333679) to be reduced by one-half
Area under plasma concentration-time curve [AUC(0-t)] of selexipag and ACT-333679 | From predose until 72 hours postdose for each treatment period
  AUC(0-t) is the area under plasma concentration-time curves for selexipag and its metabolite (ACT-333679), calculated from zero to time t of the last measured concentration above the limit of quantification
Incidence of treatment-emergent adverse events and serious adverse events | From first administration of selexipag (Day 1 Period 1) to end of study (Day 4, Period 2)
  A treatment-emergent AE is any AE temporally associated with the use of a study treatment, whether or not considered related to the study treatment, including any abnormalities in ECG parameters, vital signs or laboratory tests
Incidence of safety events of interest | From first administration of selexipag (Day 1 Period 1) to end of study (Day 4, Period 2)
  Events of interest include any abnormalities in ECG, vital signs or laboratory test results

CONTACTS AND LOCATIONS:
Overall Officials: Margaux Boehler — Actelion

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boehler M, Bruderer S, Ulc I, Dingemanse J. Biocomparison Study of Adult and Paediatric Dose Strengths of the Prostacyclin Receptor Agonist Selexipag. Eur J Drug Metab Pharmacokinet. 2018 Feb;43(1):115-120. doi: 10.1007/s13318-017-0424-z. PMID 28639216